CLINICAL TRIAL: NCT05227391
Title: Live Birth After Letrozole-stimulated Cycles Versus Hormone Replacement Treatment Cycles for the First Frozen Embryo Transfer in Women With PCOS: a Randomized Controlled Trial
Brief Title: Live Birth After Letrozole-stimulated Cycles Versus Hormone Replacement Treatment Cycles for the First Frozen Embryo Transfer in Women With PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2022001
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: PCOS
MeSH Terms: interventions — Letrozole; Estradiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole-stimulated group (Experimental)
  Interventions: Procedure: Oral Letrozole
- Hormone replacement treatment group (Active Comparator)
  Interventions: Procedure: Oral estradiol valerate

INTERVENTIONS:
Procedure: Oral Letrozole — Oral Letrozole at a dose of 2.5mg daily will be started on days 3-5 of the menstrual cycle and will be continued for 5 days.
  Arms: Letrozole-stimulated group
Procedure: Oral estradiol valerate — Oral estradiol valerate at a dose of 3mg twice daily will be started on days 3-5 of the menstrual cycle.
  Arms: Hormone replacement treatment group

SUMMARY:
This is a multicenter randomized controlled trial comparing the efficacy and safety of two endometrial preparation protocols for the first frozen embryo transfer cycle in PCOS with whole embryo freezing. Subjects will be randomized to letrozole-stimulated group or hormone replacement treatment group in their first frozen embryo transfer cycle, and their pregnancy and perinatal outcomes during this cycle will be followed up and analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1. women diagnosed with PCOS according to modified Rotterdam criteria;
* 2. Women who are participating in their first cycle of IVF or ICSI.
* 3. Women whose IVF/ICSI ovarian stimulation protocol was either GnRH antagonist protocol or long agonist protocol.
* 4. Women with whole embryos freezing.
* 5. Women aged 20 to 38 years old;
* 6. Women BMI 18 kg/m2 to 30 kg/m2
* 7. Women with at least one good-quality embryo suitable for transfer, including day 3 cleavage stage embryo with grade 7CI /8CI and day 5 or day 6 blastocyst with grade 4BB or higher.

Exclusion Criteria:

* 1. Women who has a history of recurrent spontaneous abortion.
* 2. Women with unilateral/bilateral oophorectomy.
* 3. Women with untreated Hydrosalpinx.
* 4. Women with a uterine cavity abnormality, such as a uterine congenital malformation, untreated uterine septum (except shallow uterine septum), adenomyosis, submucous myoma, or moderate to severe intrauterine adhesions.
* 5. Women with uncontrolled diabetes mellitus, thyroid disease and hypertension.
* 6. Women who are indicated and planned to undergo preimplantation genetic test (PGT).

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1078 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 11 months
  Number of women with live birth/ number of women randomized to the specific group. Live birth is defined as the delivery of any viable infant at 28 weeks or more of gestation.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 2 months
  Number of women with clinical pregnancy /number of women randomized to the specific group. Clinical pregnancy was defined as the presence of at least one gestational sac in the uterine cavity on ultrasound at about 28 days after embryo transfer.
Biochemical pregnancy rate | 1.5 months
  Number of women with biochemical pregnancy /number of women randomized to the specific group. Biochemical pregnancy was defined as a human chorionic gonadotropin level of more than 10 milli-International unit (mIU) per milliliter (ml) as measured at about 14 days after embryo transfer.
Miscarriage rate | 9 months
  Number of women with miscarrage / number of women with clinical pregnancy. Miscarriage refers to a complete spontaneous abortion or a nonviable pregnancy before 28 weeks of gestation.
Cycle cancellation rate | 1 month
  Number of women who initiated endometrial preparation without embryos transfer / number of women randomized to the specific group.
Birth weight | 11 months
  Weight of newborns at delivery.
Incidence of obstetric and perinatal complications | 11 months
  Number of pregnancies with complications / number of clinical pregnancies.
Incidence of neonatal complications | 11 months
  Number of live births with neonatal complications / number of live births.
Ectopic pregnancy rate | 2 months
  Number of women with ectopic pregnancy /number of women randomized to the specific group. Ectopic pregnancy will be defined as implantation outside the uterine cavity, as confirmed by sonography or laparoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-Xiangya, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data collected during the trial will be shared after deidentification upon request.
  Study protocol, Statistical analysis plan, informed consent forms, and clinical study report will be available upon request.
  Data will be available from 3 months following first publication and ending 5 years after the study has been concluded.
  Individual participant data will be shared with researches who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from 3 months following first publication and ending 5 years after the study has been concluded.
Access Criteria: Individual participant data will be shared with researches who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee.

REFERENCES:
- [Derived] Wang X, Li Y, Zhang C, Feng YR, Deng B, Zhang S, Ma Y, Wu Y, Lin G, Gong F. Live birth after letrozole-stimulated cycles versus hormone replacement treatment cycles for the first frozen embryo transfer in women with polycystic ovary syndrome: protocol for a multicentre randomised controlled trial. BMJ Open. 2023 Aug 17;13(8):e072021. doi: 10.1136/bmjopen-2023-072021. PMID 37591656